CLINICAL TRIAL: NCT06333314
Title: Dostarlimab as First-line Treatment for Patients With dMMR/MSI (Non-colorectal/Non-endometrial) Locally Advanced or Metastatic Cancer: a Randomized Phase 2 Trial (Cohort Pan-MSI ACSE) With Crossover in the Standard Arm at Progression
Brief Title: Dostarlimab for Locally Advanced or Metastatic Cancer (Non-colorectal/Non-endometrial) With Tumor dMMR/MSI
Acronym: Pan-MSI-ACSE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: National Cancer Institute, France (Other Government); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-IMM-2302
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Adenocarcinoma; Ampulla of Vater Carcinoma; Adrenocortical Carcinoma; Neuroendocrine Carcinoma; Soft Tissue Sarcoma; Small Bowel Adenocarcinoma; Duodenum Adenocarcinoma; Gastric Adenocarcinoma
Keywords: Immunotherapy; locally advanced or metastatic cancer; dMMR/MSI (non-colorectal/non-endometrial) cancer
MeSH Terms: conditions — Adrenocortical Carcinoma; Carcinoma, Neuroendocrine; Sarcoma; Neoplasm Metastasis; Neoplasms | interventions — dostarlimab; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, multicenter, comparative phase II trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dostarlimab (Experimental): Patient will receive dostarlimab intravenously 500 mg every 3 weeks for 4 cycles followed by 1000 mg every 6 weeks for all cycles thereafter until disease progression, unacceptable toxicity, death, investigator's decision, patient's decision or for a maximum of 24 months.
  Interventions: Drug: Dostarlimab
- Standard of care (Active Comparator): Patients will receive the standard of care chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Dostarlimab — Anti-PD-1 monoclonal antibody
  Arms: Dostarlimab
Drug: Chemotherapy — * mFOLFOX6 or FOLFIRI or XELOX regimen
  * FOLFOX or XELOX or TFOX regimen
  * FOLFIRINOX or gemcitabine-nab-paclitaxel or gemcitabine monotherapy.
  * Cisplatin and gemcitabine cisplatin or CAPOX or mFOLFOX6.
  * Etoposide-cisplatin-doxorubicin or mitotane
  * Cisplatin and gemcitabine or carboplatin and paclitaxel
  * Etoposide-cisplatin or etoposide-carboplatin
  * Doxorubicin and ifosfamide or doxorubicin monotherapy or doxorubicin and trabectedin.
  Arms: Standard of care

SUMMARY:
The goal of this open-label randomized, multicenter, comparative phase II trial is to evaluate the efficacy of the immunotherapy, dostarlimab, as first-line treatment for deficient mismatch repair (dMMR)/microsatellite instability (MSI) non-resectable metastatic or locally advanced non-colorectal and non-endometrial cancers compared to the standard of care chemotherapy.

Adult patients (aged ≥18 years) with histologically confirmed dMMR/MSI duodenum and small bowel adenocarcinoma, gastric and oeso-gastric junction (OGJ) adenocarcinoma with combined positive score (CPS)<5, pancreatic adenocarcinoma, ampulla of vater adenocarcinoma, adrenocortical carcinoma, carcinoma of unknown primary site, neuroendocrine carcinoma (Grade3) all primary, and soft tissue sarcoma (except Gastro-Intestinal Stromal Tumor) will be included in this study. They will be randomized and treated with either dostarlimab (experimental arm A), or chemotherapy (control arm B).

Patients with documented disease progression following the first line chemotherapy (Arm B) may be eligible for crossover to be treated with dostarlimab, with the same schedule as arm A.

DETAILED DESCRIPTION:
Following signature of the informed consent form, patients will enter the pre-inclusion period (maximum 28 days prior to start of treatment) during which all examinations required to assess their eligibility will be performed, including dMMR/MSI status, demographic data collection, tumor evaluation, and clinical and laboratory evaluations. A centralized confirmation of MMR/MSI status by immunohistochemistry (IHC) or next-generation sequencing (NGS)/polymerase chain reaction (PCR) is mandatory to include the patient.

Patients will be randomized 1:1 to receive either dostarlimab intravenously 500 mg every 3 weeks for 4 cycles followed by 1000 mg every 6 weeks for all cycles thereafter (experimental arm A) or chemotherapy (control arm B) as per standard of care (SOC) until disease progression, unacceptable toxicity, death, investigator's decision, withdrawal of consent or for a maximum of 24 months.

Randomization will be stratified by:

* Primary tumor (Duodenum and Small Bowel/Gastric/OGJ vs Pancreas/ Ampulla of Vater vs Other),
* Age (<70 years vs ≥70 years)
* Stage: Locally advanced vs Metastatic.

Patients randomized to Arm B may be eligible to participate in the crossover phase after documentation of disease progression by investigator evaluation according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1). Crossover patients may then be treated with dostarlimab for up to 2 years, according to the schedule defined for experimental arm A. These patients may not initiate treatment with dostarlimab any earlier than 28 days after their last dose of chemotherapy (washout period) regardless of the time of progression. Patients who discontinue dostarlimab treatment after crossover will enter the follow-up phase until the last follow-up visit of the last randomized patient. Crossover is optional and is at the discretion of the investigator (with coordinating investigator's agreement).

In both arms, tumor evaluation will be done by local investigator at inclusion and post-randomization visits as follow:

* Treatment period: every 6 weeks (+/- 7 days) for the first year then every 12 weeks (+/- 7 days) for the second year.
* Follow-up period: every 16 weeks (+/- 7 days) up to one year after the last follow-up of the last randomized patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent form prior any trial specific procedures. -
2. 18 years or older patients.
3. Documented locally advanced or metastatic disease with no previous systemic anti-cancer treatment in these settings and not suitable for complete surgical resection.
4. Histologically proven, dMMR/MSI-H solid tumors that are not colorectal or endometrial cancers and including one of the following: duodenum and small bowel adenocarcinoma, gastric and oeso-gastric junction adenocarcinoma with CPS<5, pancreatic adenocarcinoma, ampulla of Vater adenocarcinoma, adrenocortical carcinoma, carcinoma of unknown primary site, neuroendocrine carcinoma (Grade 3) all primary, and soft tissue sarcoma except Gastro-Intestinal Stromal Tumor (GIST).
5. If patient received adjuvant therapy for non-metastatic disease, this therapy should be completed more than 6 months before the diagnosis of metastatic or recurrent disease.
6. Availability of minimum 1 block of tumor tissue or 20 slides (archival (<2 years) or fresh biopsy specimen of primary and or metastasis) for centralized confirmation of MMR/MSI status by IHC or NGS/PCR, and for Translational Research.
7. Patients with dMMR/MSI tumor analyzed by IHC, PCR (for Gastric and OGJ adenocarcinoma, and duodenum and small bowel adenocarcinoma only), and/or NGS at the recruiting center should be confirmed by central review within 24h (every anonymized patient analysis reporting will be provided for central review). Patients should not be included in the study until the dMMR/MSI status is confirmed by the review committee.

   NB: In case of ambiguous result of IHC (lack of positive internal control, heterogeneous loss of MMR protein expression, ambiguous loss of only one protein including HMSH6 and PMS2), the MSI-H status will be assessed by PCR or NGS for gastric and OGJ adenocarcinoma, and duodenum and small bowel adenocarcinoma, and by NGS for other primary. Based on IHC and PCR or NGS results (NGS will be centrally performed in this case ), the sponsor will decide if inclusion is possible;
8. Presence of at least one measurable lesion within 28 days before the start of treatment according to RECIST v1.1.
9. Eastern Cooperative Oncology Group Performance status (ECOG PS) 0-1.
10. Haematological status: absolute neutrophil count (ANC) ≥1.5 x 10⁹/L; platelets ≥100 x 10⁹/L; haemoglobin ≥9 g/dL.
11. Adequate renal function: serum creatinine level <120 µM, or clearance >50 ml/min (Modification of the Diet in Renal Disease [MDRD] or Cockcroft and Gault).
12. Adequate liver function: serum bilirubin ≤1.5 x upper normal limit (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 x ULN, unless liver metastases are present, in which case they must be ≤ 5× ULN.
13. For patients not taking warfarin: International normalised ratio (INR) <1.5 or prothrombin time (PT) <1.5 x ULN and either partial thromboplastin time (PTT) or activated PTT (aPTT) <1.5 x ULN. Participants taking warfarin may be included on a stable dose with a therapeutic INR <3.5.
14. Women of childbearing potential must have a negative serum pregnancy test performed within 72 hours before the date of randomization.
15. Men, and women of childbearing potential must agree to use adequate contraception for the duration of trial participation and for 4 months after the last dose of dostarlimab (used in first line or at crossover) or for at least 6 months after the last administration of the chemotherapy agent(s) used in the control arm if no crossover with dostarlimab (according to the current version of the summary of product characteristics (SmPC) of each chemotherapy agent). Men must also agree to not donate sperm and women must agree to not donate oocytes during the specified period.
16. Registration in a National Health Care System.
17. Patient is willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study.

Exclusion Criteria:

1. Colorectal and endometrial cancer and all primary tumor not listed in inclusion criterion #4.
2. Previous exposure to anti-PD-1 or PD-L1 or anti-CTL-4 antibodies or treatment with immunotherapy.
3. Previous exposure to any investigational drug within 4 weeks (6 weeks for monoclonal antibodies) before the first dose in the study.
4. Previous exposure to any systemic anti-cancer therapy or radiation therapy for the cancer for which the patient is being enrolled.
5. Active autoimmune disease: Active autoimmune disease requiring systemic treatment in the past 2 years (excluding replacement therapy) or any history of interstitial lung disease (patients with ancient auto-immune disease with stable endocrine oral substitution are eligible).
6. Uncontrolled central nervous system metastases or carcinomatous meningitis or other concurrent illness or ongoing or active infections.
7. Patients with HER2-positive gastric carcinoma.
8. Other serious and uncontrolled non-malignant disease or is considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active infection requiring systemic therapy. Specific examples include, but are not limited to, active, non-infectious pneumonitis; uncontrolled ventricular arrhythmia; recent (within 90 days) myocardial infarction; uncontrolled major seizure disorder; unstable spinal cord compression; superior vena cava syndrome; or any psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
9. Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
10. Has received treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to the first dose of adjuvant treatment or is required to receive systemic immunosuppressive medications during the study. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

    Note 1: Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled into the study after approval of the Medical Contact.

    Note 2: patients are permitted the use of topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Adrenal replacement steroid doses including doses >10 mg daily prednisone are permitted. A brief (less than 3 weeks) course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by a contact allergen) is permitted.
11. Other concomitant or previous malignancy other than the disease under study, except as noted below:

    i. adequately treated in-situ carcinoma of the uterine cervix, ii. basal or squamous cell carcinoma of the skin, iii. cancer from which the patients was in complete remission for >2 years.
12. Known Human Immunodeficiency Virus (HIV) infection.
13. Received live vaccine within 14 days.
14. Patient has documented presence of HBsAg [or HBcAb] at pre-inclusion visit or within 3 months prior to first dose of study intervention.

    Participant has a positive hepatitis C virus (HCV) antibody test result at pre-inclusion visit or within 3 months prior to first dose of study intervention. Note: Participants with a positive HCV antibody test result due to prior resolved disease can be enrolled, only if a confirmatory negative HCV RNA test is obtained.

    Participant has a positive HCV RNA test result at pre-inclusion visit or within 3 months prior to first dose of study intervention. Note: The HCV RNA test is optional and participants with negative HCV antibody test are not required to undergo HCV RNA testing as well
15. Known prior severe hypersensitivity to investigational product or any component in its formulation.
16. Pregnant or breast feeding women.
17. Participation in another clinical trial within 30 days prior to the first study treatment administration or concomitantly with the trial.
18. Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
19. Person deprived of their liberty or under protective custody or guardianship.

Patient randomized to receive SOC (Arm B) may crossover to receive dostarlimab (Arm A) in case of documented progressive disease according to RECIST v1.1.

Inclusion and exclusion are the same for the crossover except for the inclusion criteria #3 and #4.

The criterion #3 for crossover is: Patient included in the protocol and randomized in the arm "standard of care" with documented progressive disease by RECIST v1.1 on standard of care (defined in the protocol).

The criterion #4 for crossover is: Previous exposure to chemotherapy for locally advanced or metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From randomization until disease progression or death from any cause, up to 3 years.
  The progression-free survival is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.

SECONDARY OUTCOMES:
Objective Response Rate | From randomization to disease progression or death, up to 3 years
  Objective Response Rate is defined as the proportion of patients with best response of complete response (CR) or partial response (PR) according to RECIST v1.1.
Duration of response | From randomization to disease progression or death, up to 3 years
  Duration of response (DOR) will be evaluated in patients with either a complete response (CR) or partial response (PR). DOR is defined as the time from the first assessment of a CR or PR until the date of the first occurrence of progressive disease (PD) or death from any cause (if death occurred within predefined period), whichever occurs first.
Overall Survival | From randomization until death from any cause, up to 3 years
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Progression-Free Survival 2 | From randomization to disease progression or death, up to 3 years
  Progression-Free Survival 2 (PFS2) is defined as the time from randomization to second/subsequent disease progression after initiation of new anti-cancer therapy (including subsequent immune checkpoint inhibitor therapy), or death from any cause, whichever first.
Objective response rate 2 | From randomization to disease progression or death, up to 3 years
  Objective response rate after initiation of new anti-cancer therapy (ORR2) is defined as the proportion of patients with best response of CR or PR according to the investigator's judgment.
Progression-Free Survival -crossover | From randomization to disease progression or death, up to 3 years
  Progression-free survival - crossover is defined as the time from crossover initiation to disease progression after initiation of new anti-cancer therapy, or death from any cause, whichever first.
Circulating tumor DNA level | From randomization to disease progression or death, up to 3 years
  The evolution of circulating tumor DNA (ctDNA) level in patient's blood during treatment will be correlated with PFS in the overall population.
Incidence of treatment-emergent adverse events | Throughout study completion, up to 3 years
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, every 2 or 3 weeks, and at the end of treatment (up to 2 years)
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry ANDRE, MD, Principal Investigator — Hôpital Sainte Antoine - Paris - France
Locations (22):
- France (22):
  - Institut de Cancérologie de l'Ouest, Angers
  - Institut du Cancer Avignon-Provence, Avignon
  - CHU Jean Minjoz, Besançon
  - CHU Morvan, Brest
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU - Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Hôpital la Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancérologie de Lorraine, Nancy
  - Institut Mutualiste Montsouris, Paris
  - CHU de Bordeaux - Hôpital Haut -Lèvêque, Pessac
  - CHU de Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - CHU de Rouen, Rouen
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - CHU de Toulouse Hôpital Rangueil, Toulouse
  - Gustave Roussy Grand Paris, Villejuif
  - Hôpital Saint-Antoine, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No